CLINICAL TRIAL: NCT03156439
Title: Evaluation of the Bioavailability, Safety, and Tolerability of BIS-001 ER Following Multiple Dose Administration in Healthy Subjects
Brief Title: Bioavailability, Safety, and Tolerability of BIS-001 ER
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Collaborators: Melbourne Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BNI-01-1b
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Epilepsy, Complex Partial
MeSH Terms: conditions — Epilepsy, Complex Partial | interventions — huperzine A

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BIS-001 ER (Experimental): The subjects will be dosed twice daily (BID); in an on-site setting at dose initiation and at times of dose escalation to evaluate safety, and for specimen collection for routine laboratory and pharmacokinetic analysis. Subjects will be discharged and compliance of BID dosing will be monitored via twice daily phone calls by site staff. The initial dose will be 0.5mg BID with a dose escalation every 2-3 days until a maximum tolerated dose is observed or a maximum of 2.5mg BID dose is obtained.
  Interventions: Drug: BIS-001 ER

INTERVENTIONS:
Drug: BIS-001 ER — BIS-001 ER is an extended release formulation of the nutritional supplement Huperzine A.
  Other Names: Huperzine A

SUMMARY:
This study investigates the safety, tolerability, and pharmacokinetics of BIS-001 ER in healthy volunteers. Subjects will be dosed twice daily, with a dose escalation occurring every 2-3 days until a maximum dose of 5mg per day is reached.

ELIGIBILITY:
Inclusion Criteria:

1. Speak English with sufficient proficiency to read and comprehend the Informed Consent document, and to communicate with study staff.
2. Be able to consent to participate by signing the Informed Consent document after a full explanation of the nature and purpose of this study.
3. Have signed the Informed Consent before any study-specific procedures are performed
4. Be males or females between 18 - 45 years of age.
5. Have a negative urinary pregnancy test upon admission to the site on Day 1
6. Be in good general health in the judgment of the Principal Investigator based upon medical history, physical examination, standard 12-lead electrocardiogram (ECG), and clinical laboratory evaluations obtained within the two weeks prior to enrollment.
7. Be able to comply with all study-specified procedures.
8. Weight between 40 and 100 kg

Exclusion Criteria:

1. Has taken Huperzine A.
2. Is planning to become pregnant or impregnate spouse, not using an acceptable method of birth control (defined as use of double-barrier birth control methods, use of oral contraceptives, or surgical sterilization), pregnant or nursing
3. Has a pre-existing medical condition (including an existing progressive or degenerative neurological disorder) or takes medications that, in the Principal Investigator's opinion, could interfere with the subject's suitability for participation in the study.
4. Has a history or evidence of significant psychiatric disturbance or illness, including alcohol or drug abuse within the past 2 years, or symptoms of psychosis (hallucinations, delusions) in the last 5 years.
5. Has had any clinical laboratory abnormalities within the past two months, prior to screening, considered of clinical significance by the Principal Investigator
6. Is on concomitant therapy with non-anti-epileptic drugs (AEDs) that are cholinergic.
7. Has participated in any clinical investigational drug or device study within four weeks prior to study entry.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Maximum serum concentration; Cmax | 16 Weeks
  Bioavailability/Pharmacokinetic Assessments
Area under the curve; AUC | 16 Weeks
  Bioavailability/Pharmacokinetic Assessments
Time of maximum serum concentration; Tmax | 16 Weeks
  Bioavailability/Pharmacokinetic Assessments
Half-life; t1/2 | 16 Weeks
  Bioavailability/Pharmacokinetic Assessments
Terminal elimination | 16 Weeks
  Bioavailability/Pharmacokinetic Assessments
Clearance | 16 Weeks
  Bioavailability/Pharmacokinetic Assessments
Volume of distribution | 16 Weeks
  Bioavailability/Pharmacokinetic Assessments
Mean residence time | 16 Weeks
  Bioavailability/Pharmacokinetic Assessments

SECONDARY OUTCOMES:
Safety and Tolerability Assessments - Adverse Events | 16 Weeks
  Adverse events will be defined, documented, evaluated (mild/moderate/severe/life threatening; serious/non-serious; expected/unexpected; causally related to study drug or not) and reported according to all applicable institutional and governmental requirements and guidance.
Safety and Tolerability Assessments - Vital Signs | 16 Weeks
  Vital signs (e.g. blood pressure) will be monitored through the first 8 hrs after drug administration, as well as at Baseline and pre-dose.
Safety and Tolerability Assessments - Neurological Evaluation | 16 Weeks
  A standard neurological examination will be performed according to the study-specific timeline. Clinically significant new or worsened abnormalities as compared to baseline findings will have to be reported as AEs.
Safety and Tolerability Assessments - Physical Evaluation | 16 Weeks
  A standard physical examination will be performed according to the study-specific timeline. Clinically significant new or worsened abnormalities as compared to baseline findings will have to be reported as AEs.
Safety and Tolerability Assessments - ECG Evaluation | 16 Weeks
  A standard 12-lead ECG in a supine position after a 5-minute rest will be performed according to the study-specific timeline.
  The Investigator will determine whether the results of the ECG are normal or abnormal and assess the clinical significance of any abnormality. ECG tracings will be reviewed by a cardiologist if required.
Safety and Tolerability Assessments - Clinical Laboratory Studies: Hematology | 16 Weeks
  Laboratory assessments will be conducted using standard methods.
Safety and Tolerability Assessments - Clinical Laboratory Studies: Biochemistry | 16 Weeks
  Laboratory assessments will be conducted using standard methods.
Safety and Tolerability Assessments - Clinical Laboratory Studies: Urinalysis | 16 Weeks
  Laboratory assessments will be conducted using standard methods.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Collins, Study Chair — President and CEO
Locations (1):
- The Royal Melbourne Hospital, Parkville, Victoria, Australia